CLINICAL TRIAL: NCT04756154
Title: Assessment of the Antimicrobial Efficacy of 3M™ SoluPrep™ Preoperative Skin Preparation Against Resident Human Skin Flora on the Inguinal Region
Brief Title: Efficacy Study of Patient Preoperative Preps In-vivo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EM-05-014624
Record Dates: First submitted 2021-01-20; First posted 2021-02-16 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Surgical Skin Preparation
MeSH Terms: interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CHG/IPA Surgical skin preparation (Experimental): Apply topically to the inguinal region for 2 minutes
  Interventions: Drug: CHG/IPA Surgical skin preparation
- CHG/IPA Film-Forming Surgical skin preparation (Active Comparator): Apply topically to the inguinal region for 2 minutes
  Interventions: Drug: CHG/IPA Surgical skin preparation
- Normal saline (Placebo Comparator): Apply topically to the inguinal region for 2 minutes
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: CHG/IPA Surgical skin preparation — Apply topically to the inguinal region for 2 minutes
  Other Names: 2% CHG/70% IPA
  Arms: CHG/IPA Film-Forming Surgical skin preparation; CHG/IPA Surgical skin preparation
Drug: Normal saline — Apply topically to the inguinal region for 2 minutes
  Other Names: 0.9% sodium chloride
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine the antimicrobial efficacy of an investigational CHG/IPA prep on skin flora of the inguinal regions of human subjects.

DETAILED DESCRIPTION:
Non-inferiority of the investigational product to the FDA-approved active control for log10/cm2 recovery of skin flora relative to Treatment Day baseline log10/cm2 on the inguinal region at 10 minutes following application. Non-inferiority is based on a non-inferiority margin of 0.5 log10/cm2.

Superiority of the active products to the negative control for log10/cm2 recovery of skin flora relative to Treatment Day baseline log10/cm2 on the inguinal region at 10 minutes following application. A superiority margin of 1.2 log10/cm2 is used.

Number of observations for which the log10/cm2 recovery of skin flora on the inguinal region at 6 hours following application of the study products is higher than treatment day log10/cm2 baseline skin flora.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race
* Subjects in good health
* Minimum skin flora baseline requirements on inguinal region

Exclusion Criteria:

* Any tattoos, scars, breaks in the skin, or any form of dermatitis, or other skin disorders (including acne) on the applicable test area
* Topical antimicrobial exposure within 14 days prior to screening and treatment days
* Use of systemic or topical antibiotics, steroid medications, or any other products known to affect the normal microbial flora of the skin within 14 days prior to screening and treatment days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad H Bashir, MD, CCRP, Principal Investigator — Microbac
Locations (1):
- Microbac Laboratories, Inc, Sterling, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomized, paired-comparison design where each subject received two of the planned treatments, one on the left side and one on the right. Each subject provided two inguinal test sites, left and right. 154 subjects were randomized for the inguinal region resulting in 308 applications of test products.
Units Other Than Participants: Test sites on skin
Period: Overall Study
Arm/Group | CHG/IPA Surgical Skin Preparation | CHG/IPA Film-Forming Surgical Skin Preparation | Normal Saline
Started | 135; 135 Test sites on skin | 135; 135 Test sites on skin | 38; 38 Test sites on skin
Completed | 104; 104 Test sites on skin | 106; 106 Test sites on skin | 31; 31 Test sites on skin
Not Completed | 31; 31 Test sites on skin | 29; 29 Test sites on skin | 7; 7 Test sites on skin
Not completed — Did not meet treatment day baseline | 30 | 28 | 7
Not completed — Did not return for final sample collection | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with average treatment day baseline counts of greater than or equal to 5.00 log10 CFU/cm^2 bilaterally on the inguinal region were included in the analysis.
Units Other Than Participants: Test sites on skin
Groups:
- Total: Total of all reporting groups
Arm/Group | CHG/IPA Surgical Skin Preparation | CHG/IPA Film-Forming Surgical Skin Preparation | Normal Saline | Total
Number analyzed (Participants) | 135 | 135 | 38 | 154
Number analyzed (Test sites on skin) | 135 | 135 | 38 | 308
Age, Customized [Number; unit: Test sites on skin]
  Between 18-65 years | 126 | 126 | 38 | 290
  > 65 years | 9 | 9 | 0 | 18
Sex/Gender, Customized [Number; unit: Test sites on skin]
  Female | 62 | 62 | 16 | 140
  Male | 73 | 73 | 22 | 168
Race/Ethnicity, Customized [Number; unit: Test sites on skin]
  American Indian or Alaska Native | 2 | 2 | 0 | 4
  Asian | 61 | 64 | 13 | 138
  Black or African American | 18 | 21 | 5 | 44
  Native Hawaiian | 1 | 2 | 1 | 4
  White | 49 | 43 | 18 | 110
  Other | 4 | 3 | 1 | 8
Region of Enrollment [Number; unit: Test sites on skin]
  United States | 135 | 135 | 38 | 308

OUTCOME MEASURES:

1. Primary Outcome: Log Change (Reduction) in Skin Flora on the Inguinal Region at 10 Minutes
Description: Immediate efficacy endpoint which is defined as the average treatment effect (ATE) log10 CFU/cm2 of skin flora on the inguinal region at 10 minutes following application of the study products relative to the treatment day baseline skin flora
Time Frame: 10 minutes
Population: The primary analysis data set used a modified intent-to-treat population. Subjects were excluded who did not meet the treatment day baseline requirements of 5.00 log10/cm^2 on the inguinal test site. The number treatment arm-specific test sites is equal to the number of participants.
Measure: Mean (Standard Deviation); unit: Log10 CFU/cm^2
Groups:
- CHG/IPA Film-Forming Surgical Skin Preparation:; Normal Saline: Apply topically to the inguinal region for 2 minutes
Arm/Group | CHG/IPA Surgical Skin Preparation | CHG/IPA Film-Forming Surgical Skin Preparation: | Normal Saline
Number analyzed (Participants) | 106 | 104 | 31
Log10 CFU/cm^2 | 3.60 (0.816) | 3.61 (0.837) | 1.15 (0.411)

2. Primary Outcome: Log Change (Reduction) in Skin Flora on the Inguinal Region at 6 Hours
Description: Persistent efficacy endpoint which is a binary endpoint with success/failure, where "success" is defined as log10 CFU/cm2 of skin flora on the inguinal region at 6 hours following application of the study products being lower than the treatment day baseline skin flora
Time Frame: 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log10 CFU/cm^2
Arm/Group | CHG/IPA Surgical Skin Preparation | CHG/IPA Film-Forming Surgical Skin Preparation | Normal Saline
Number analyzed (Participants) | 106 | 104 | 31
Log10 CFU/cm^2 | 1.98 (0.806) | 2.40 (0.792) | 1.03 (0.443)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on treatment day, an average of 6-7 hours per participant. By definition, all AEs were treatment-emergent.
Arm/Group | CHG/IPA Surgical Skin Preparation | CHG/IPA Film-Forming Surgical Skin Preparation | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/135 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/135 | 0/38
Other Adverse Events (participants affected / at risk) | 0/135 | 0/135 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Combined Protocol and Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT04756154/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Detailed Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT04756154/SAP_001.pdf